CLINICAL TRIAL: NCT00151840
Title: Efficacy and Safety of IVIG-L (Human Normal Immunoglobulin for Intravenous Use)in Idiopathic Thrombocytopenic Purpura (ITP)Patients
Brief Title: Efficacy and Safety of IVIG-L in ITP Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prothya Biosolutions (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB98001
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2006-01-31 (Estimated); Status verified 2006-01

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic
Keywords: Purpura, Thrombocytopenic, Idiopathic; ITP; Immunoglobulin, Intravenous
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

INTERVENTIONS:
Drug: IVIG-L

SUMMARY:
The efficacy and safety of a liquid intravenous immunoglobulin product, IVIG-L, in patients with ITP will be assessed and compared with data obtained from literature.

DETAILED DESCRIPTION:
Sanquin has developed, in cooperation with the Finnish Red Cross Blood Transfusion Service (FRCBTS), a liquid intravenous immunoglobulin product, IVIG-L. The liquid formulation of intravenous immunoglobulin simplifies infusion, eliminates possible mistakes in the reconstitution with water for injection and reduces space requirements in storage.

In addition to donor selection and screening, several procedures have been included in the production process to improve viral safety.

In this clinical trial, the efficacy and safety of IVIG-L in patients with ITP will be assessed and compared with data obtained from literature. IVIG-L will also be studied in patients with hypogammaglobulinemia.The results from both studies will be used for an application for marketing authorisation of IVIG-L in Finland and the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic ITP with a platelet count of about 20x109/L and at high risk of bleeding
* Patients with chronic ITP with a platelet count of about 20x109/L, who have to undergo surgery
* A stable clinical situation (no activity of any other disease)
* Age at least 18 yrs
* The patient/legally acceptable representative has signed the consent form

Exclusion Criteria:

* The presence of another autoimmune disease related with thrombocytopenia such as systematic lupus erythematosus (SLE), rheumatoid arthritis (RA) or nephritis
* Patients with drug-induced thrombocytopenia or immunologic thrombocytopenia of infectious origin (in particular, Hepatitis, Epstein-Barr virus, Toxoplasma, HIV)
* Massive splenomegaly
* Treatment with any other investigational drug within 7 days before study entry or previous enrolment in this study
* Having an ongoing progressive terminal disease, including HIV infection
* Known with allergic reactions against human plasma, plasma products or intravenous immunoglobulin
* Presence of conditions predisposing for bleeding: anaemia (hemoglobin < 5.5 mmol/L), renal or urogenital disease, malignant disease (with the exception of basalioma, cervix carcinoma in situ), history of intracranial or aortic aneurysm, stroke, oeso-gastro-intestinal disorders with a bleeding potential, severe hypertension (diastole > 110 mm Hg).
* Use of corticosteroids for an acute situation within 7 days before study entry. Patients using corticosteroids prophylactically can be included
* Splenectomy in the previous two weeks
* Renal insufficiency (plasma creatinine > 115µmol/L)
* Pregnancy or lactation
* Known with insufficiency of coronary or cerebral circulation
* IgA deficiency and anti-IgA antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2001-10; Study Completion 2002-03

PRIMARY OUTCOMES:
The efficacy of IVIG-L
The safety of IVIG-L

SECONDARY OUTCOMES:
To compare data on efficacy and safety of IVIG-L with data obtained from literature

CONTACTS AND LOCATIONS:
Overall Officials: P FW Strengers, MD, Study Director — Prothya Biosolutions
Locations (6):
- Poland (6):
  - Hematology Clinic, Medical University of Bialystok, Bialystok
  - Haematology Clinic, Medical University of Gdansk, Gdansk
  - Clinic of Haematology, Medical University of Lodz, Lodz
  - Clinical of Internal Diseases and haematology with Bone marrow Transplantation Unit, Central Academic Hospital, Medical Military Academy, Warsaw
  - Institute of Haematology and Transfusiology, Warsaw
  - Haematology Clinic, Medical University of Warsaw, Warsaw